CLINICAL TRIAL: NCT06780215
Title: Efficacy of Varenicline Tartrate in Treating Frequent Premature Ventricular Contractions: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial (Var-PVC)
Brief Title: Efficacy of Varenicline Tartrate in Treating Frequent Premature Ventricular Contractions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yihan Chen (Other)
Responsible Party: Sponsor-Investigator, Yihan Chen, President, Shanghai East Hospital, Shanghai East Hospital
Organization: Shanghai East Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025YS-002; NCT06780215 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Premature Ventricular Contraction (PVC)
Keywords: Premature ventricular contractions; Varenicline; Myocardial infarction
MeSH Terms: conditions — Ventricular Premature Complexes; Myocardial Infarction | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, multicenter, randomized, double-blind, parallel-group，placebo-controlled superiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants receive placebo tablets according to the treatment group design.
  Interventions: Drug: Placebo
- Treatment Group (Experimental): Participants take varenicline tartrate tablets according to the regimen
  Interventions: Drug: Varenicline Tartrate Tablets

INTERVENTIONS:
Drug: Varenicline Tartrate Tablets — Participants in treatment group take varenicline tartrate tablets according to the following regimen:
  Days 1-3: 0.5 mg/dose, once daily. Days 4-42: 0.5 mg/dose, twice daily, taken orally at the same time each morning and evening (the dosing interval is recommended to be 12 h ± 2 h).
  Days 43-45: 0.5 mg/dose, once daily.
  Arms: Treatment Group
Drug: Placebo — Days 1-3: 1 tablet/dose, once daily. Days 4-42: 1 tablet/dose, twice daily, taken orally at the same time each morning and evening (the dosing interval is recommended to be 12 h ± 2 h).
  Days 43-45: 1 tablet/dose, once daily.
  Arms: Control Group

SUMMARY:
This is an investigator-initiated, multicenter, randomized, double-blind, placebo-controlled, parallel-group clinical trial designed to evaluate the preliminary efficacy of varenicline tartrate in patients with frequent PVCs complicated by myocardial infarction (MI). The protocol was approved by the institutional review board and ethics committee at each participating center.

Primary Efficacy Endpoint:

1) The percentage change from baseline in the 24-hour mean count of PVCs at Week 6.

Secondary Efficacy Endpoints:

1. The responder rate for PVCs at Weeks 4, 6, and 8. PVC responder: A participant is considered a responder if there is a ≥ 50% reduction from baseline in the 24-hour mean PVC count following treatment with either varenicline or placebo.
2. The incidence of NSVT from randomization through Weeks 4, 6, and 8.
3. The change from baseline in the 24-hour mean count and burden of PVCs at Weeks 4, 6, and 8.
4. The change from baseline in the 24-hour mean episodes and burden of non-sustained ventricular tachycardia (NSVT) at Weeks 4, 6, and 8.
5. The change from baseline in the Kansas City Cardiomyopathy Questionnaire (KCCQ) score at Week 6.

Pre-specified Safety Endpoints:

Primary Endpoint: The cumulative incidence of the first occurrence of malignant ventricular arrhythmias (time-to-first event), including sustained ventricular tachycardia (SVT), ventricular fibrillation (VF), or ventricular flutter (VFL), from randomization through Weeks 4, 6, and 8.

Study Population:

A total of 116 participants, aged 18-80 years, with frequent PVCs wil be enrolled. Prior to enrollment, participants must have stable cardiac conditions and must have received standard treatment for acute or chronic coronary syndrome as recommended by the relevant guidelines, including sustained-release metoprolol succinate. Following preliminary screening, participants will undergo 72-hour continuous three-lead AECG monitoring (baseline data) to assess the baseline PVC frequency. Eligibility for inclusion will be determined based on the monitoring data. Eligible participants will then be randomized in a 1:1 ratio (Day 0) to either the treatment group (varenicline tartrate tablets) or the placebo group.

Treatment Protocol:

All participants will receive sustained-release metoprolol succinate as part of the standard treatment, in accordance with clinical guidelines. The dose will remain stable throughout the study, unless adjustments are required for patient safety. Other standard treatments recommended by the guidelines, aside from sustained-release metoprolol succinate, will be optimized according to the clinical guidelines throughout the study.

Randomization and Stratification:

A total of 116 participants will be enrolled and randomized to either the treatment or placebo group, with 58 participants in each group. Stratification will be based on left ventricular ejection fraction (LVEF ≥ 50% vs. LVEF < 50%).

Treatment Regimen:

Treatment Group (Varenicline Tartrate 0.5 mg/tablet): Participants will receive the following regimen:

Days 1-3: 0.5 mg once daily. Days 4-42: 0.5 mg twice daily, taken at the same times each day (recommended interval 12 hours ± 2 hours).

Days 43-45: 0.5 mg once daily.

Placebo Group: Participants will receive placebo tablets according to the same regimen as the treatment group:

Days 1-3: 1 tablet once daily. Days 4-42: 1 tablet twice daily, taken at the same times each day (recommended interval 12 hours ± 2 hours).

Days 43-45: 1 tablet once daily. Statistical Analysis General Principles

1. Continuous (quantitative) variables: Summarized with n, mean, standard deviation, median, interquartile range, minimum, and maximum.
2. Categorical (count) variables: Presented as n (%). Unless otherwise specified, percentages will be calculated using the number of participants in the relevant analysis population as the denominator.

Efficacy Analysis

1） Primary endpoint: The between-group difference will be assessed by estimating the mean difference in the percentage reduction from baseline in the 24-hour mean PVC count at Week 6, with 95% confidence intervals (CIs).

Secondary endpoints: Two key secondary efficacy end points will be formally tested using a fixed-sequence (hierarchical) procedure.

Key Secondary End Point 1: The responder rate for PVCs at Week 6. Key Secondary End Point 2: The incidence of NSVT at Week 6. All other secondary efficacy endpoints will be summarized descriptively. Safety Analysis The cumulative incidence of malignant ventricular arrhythmias will be estimated using Kaplan-Meier survival curves, with differences between groups compared using the Cox proportional hazards model (reporting the hazard ratio [HR] and 95% CI). If no events occur in either group or if the number of events is too low, only the number of events and their percentages will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years old (inclusive).
2. Premature ventricular contractions of ≥1000 times/average 24-hour revealed by screening (72-hour Holter monitoring).
3. Definite diagnosis of myocardial infarction for more than 4 weeks, with NYHA Class I-II.
4. Maintained on Metoprolol Succinate Sustained-release Tablets. (If other types of beta-blocker therapy were being used before screening, they must be replaced with Metoprolol Succinate Sustained-release Tablets.)
5. Understand and comply with the study procedures and methods, and sign the informed consent form.

Exclusion Criteria:

1. Myocardial infarction occurring within 4 weeks.
2. NYHA Class III-IV.
3. Use of amiodarone within 1 month before screening.
4. Use of antiarrhythmic drugs, or traditional Chinese medicine, Chinese patent medicine for arrhythmia other than amiodarone within 1 week prior to screening.
5. Sustained ventricular tachycardia, ventricular flutter, or ventricular fibrillation detected during screening (non-sustained ventricular tachycardia does not need to be excluded).
6. Sick sinus syndrome without pacemaker implantation, II-III degree atrioventricular block, or bundle branch block bilateral.
7. Moderate to severe bronchial asthma or severe chronic obstructive pulmonary disease.
8. Severe renal impairment (eGFR less than 30 mL/min/1.73 m²).
9. Hyperthyroidism.
10. Severe sequelae of stroke.
11. Epilepsy, schizophrenia, or depression.
12. Pregnant or breastfeeding women, or those with a positive blood pregnancy test result before randomization.
13. Combined cancer or other diseases, with an expected life expectancy of less than 1 year.
14. Perioperative period of cardiothoracic surgery (1 week before surgery to 2 weeks after surgery).
15. Severe electrolyte disturbance.
16. Digitalis poisoning.
17. Known hypersensitivity to varenicline tartrate tablets or their excipients.
18. History of smoking and cessation for less than 1 year.
19. Individuals taking varenicline tartrate tablets for smoking cessation.
20. Currently participating in other clinical studies.
21. Other conditions making the subjects unsuitable for enrollment as determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in the average 24-hour count of premature ventricular contractions | Week 6

SECONDARY OUTCOMES:
The responder rate for premature ventricular contractions (PVCs) . | At Weeks 4, 6, and 8.
  PVC responder: A participant is considered a responder if there is a ≥ 50% reduction from baseline in the 24-hour mean PVC count following treatment with either varenicline or placebo.
The incidence of non-sustained ventricular tachycardia (NSVT). | At Weeks 4, 6, and 8.
  If the 72-hour ECG monitoring shows a non-zero value for the number of NSVT episodes, it will be considered as "occurrence." If the number is zero, it will be considered as "non-occurrence." The incidence of NSVT at Weeks 4, 6, and 8 will be calculated by dividing the number of participants with NSVT episodes recorded by the 72-hour AECG monitoring by the total number of participants in each group, and then multiplying by 100%.
Changes from baseline in the average 24-hour count and burden of premature ventricular contractions | Weeks 4, 6, and 8
Changes from baseline in the average 24-hour number of episodes and burden of non-sustained ventricular tachycardia | Weeks 4, 6, and 8
Change from baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Week 6
  The KCCQ score ranges from 0 to 100, with higher scores indicating better outcomes.

OTHER OUTCOMES:
Safety End Points: The cumulative incidence of the first occurrence of malignant ventricular arrhythmias (time-to-first event) , including sustained ventricular tachycardia (SVT), ventricular fibrillation (VF), or ventricular flutter (VFL). | From randomization through Weeks 4, 6, and 8.
  The malignant ventricular arrhythmia events will be adjudicated by the Central Adjudication Committee (CEC) based on planned 72-hour continuous ambulatory electrocardiography (AECG) monitoring and unplanned clinical evidence, including emergency or inpatient 12-lead ECG, bedside monitoring or telemetry ECG, implantable cardioverter defibrillator (ICD) records, or cardiopulmonary resuscitation (CPR) records, using a standardized approach. An event will be counted if any of these criteria are met; each participant will be counted for a maximum of one event. The event time will be taken as the earliest verifiable evidence. The analysis will be based on the risk set starting from randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No